CLINICAL TRIAL: NCT03526211
Title: Study of Feasibility and Safety of Functional Electrical Stimulation (FES) Cycling in Intensive Care Unit Patients
Brief Title: Safety Evaluation of Functional Electrical Stimulation (FES) Cycling in Intensive Care Unit Patients
Acronym: FES Cycling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire de Physique ENS de Lyon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18CH005; 2018-A00541-54 (Other: ANSM)
Record Dates: First submitted 2018-03-28; First posted 2018-05-16 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-06

CONDITIONS: Muscle Weakness
Keywords: Intensive care unit acquired muscle weakness; Cycloergometer; Neuromuscular electrical stimulation; FES Cycling
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients with FES Cycling
  Interventions: Device: FES cycling

INTERVENTIONS:
Device: FES cycling — On the patient, three pairs of electrodes will be applied on tibial hamstring, quadriceps and gluteal muscles of each lower limb. Cycloergometer will be installed in passive mode. Then, optimal stimulation intensity for each muscle will be defined. During twenty minutes, neuromuscular electrical stimulation will generate a passive pedaling on cycloergometer.

SUMMARY:
Intensive care unit acquired muscle weakness (ICUAW), is a common disease which influence rehabilitation, extend mechanical ventilation and length of stay in intensive care unit, and affect quality of life at hospital discharge.

To prevent ICUAW, different strategies of early mobilization are recommended. But all cannot be applied in all ICU patients. Some of them benefit from heavy therapies like circulatory assistance or renal replacement therapy for example, that limit mobilization.

Cycloergometer is a tool that allows continuous passive mobilization in bedridden and even unconscious patients.

Neuromuscular electrical stimulation (NMES) is an alternative that helps preserve muscle mass and limit muscle atrophy.

Early bedside cycle exercise coupled with NMES is an interesting new approach where application of an electrical stimulation along specific motor nerves on each lower limb, generates muscles contractions and pedaling on cycloergometer.

The aim of this study is to evaluate safety and feasibility of this coupled technique called Functional Electrical Stimulation (FES) Cycling, in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Deeply sedated (Riker 1-2) patients, admitted in intensive care unit B of ST-Etienne hospital
* Without curare since 12 hours
* Normothermic or with a controlled fever (central temperature between 36 and 38°C)
* Without haemodynamic instability (mean arterial pressure > 65mmHg and < 120mmHg, systolic arterial pressure > 90mmHg and < 200mmHg, Norepinephrine < 4mg/h)
* Without respiratory instability (respiratory rate < 35/min, pulse oxymetry > 90%, inspired oxygen fraction < 60%, PaO2/FiO2 ratio > 250, Peep < 10cmH2O, with invasive mechanical ventilation)
* Without neurological instability (diastolic velocities in mean cerebral artery > 30cm/s, mean velocities > 50cm/s, pulsatility index < 1.2, intracranial pressure < 20mmhg, brain tissue oxygenation tension > 15mmHg)
* Patient whose family has given informed and written consent to the patient's participation in the study

Exclusion Criteria:

* Pregnant woman,
* Patients with peripheral nerve damage prior to or at the time of measurement
* Curarized patients (non-efficacy of neurostimulation)
* Presence of a catheter in the stimulation zone (femoral artery or vein)
* Patients with lower limb, pelvic or spine fracture
* Patients with continuous renal replacement therapy
* Patients with circulatory assistance
* Patients with wounds in electrodes placement area
* Morbidly obesity with Ideal Body Weight > 40kg/m2
* Patients with pacemaker
* Lower limb deep vein thrombosis without treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Tolerance | During the FES Cycling session (day 1)
  Number of FES Cycling sessions that must be stopped because of the presence of at least 1 following criteria (these criteria are qualitative (presence or absence) and therefore do not add up):
  * Mean arterial pressure <65mmHg or> 120mmHg,
  * Systolic blood pressure <90 mmHg or> 200 mmHg,
  * Heart rate <50 or> 130 / min
  * Occurrence of atrial or ventricular arrhythmia
  * Respiratory rate > 35 / min,
  * Pulse oxygen saturation <90%
  * Intracranial pressure > 20mmHg.
  * Mean mean arterial velocity measured by transcranial Doppler <30 cm / s

SECONDARY OUTCOMES:
Systolic blood pressure | During the FES Cycling session (day 1)
  Haemodynamic repercussions of a FES Cycling session measured by Systolic blood pressure
Haemodynamic tolerance Heart rate | During the FES Cycling session (day 1)
  Haemodynamic repercussions of a FES Cycling session measured by Heart rate
Cardiac output measured | During the FES Cycling session (day 1)
  Haemodynamic repercussions of a FES Cycling session measured by Cardiac output measured in transthoracic echocardiography
Fick equation | During the FES Cycling session (day 1)
  Haemodynamic repercussions of a FES Cycling session measured by oxygen consumption according to the Fick equation (cardiac output x (arterial content in O2 - venous content in O2))
Arterial lactates | During the FES Cycling session (day 1)
  Haemodynamic repercussions of a FES Cycling session measured Arterial lactates
Venous oxygen | During the FES Cycling session (day 1)
  Haemodynamic repercussions of a FES Cycling session measured by Venous oxygen saturation
Amine dosage | During the FES Cycling session (day 1)
  Haemodynamic repercussions of a FES Cycling session measured by Amine dosage
Respiratory tolerance Oxygen saturation | During the FES Cycling session (day 1)
  Respiratory repercussions of a FES Cycling session measured by Oxygen saturation
Respiratory tolerance | During the FES Cycling session (day 1)
  Respiratory repercussions of a FES Cycling session measured by Respiratory rate
Respiratory rate | During the FES Cycling session (day 1)
  Respiratory repercussions of a FES Cycling session measured by PaCO2 and PaO2
Diastolic cerebral artery | During the FES Cycling session (day 1)
  Neurological repercussions of a FES Cycling session measured by diastolic average cerebral artery measured by transcranial Doppler
Pulsatility index | During the FES Cycling session (day 1)
  Neurological repercussions of a FES Cycling session measured by Average of pulsatility index, measured by transcranial Doppler.
Intracranial pression | During the FES Cycling session (day 1)
  Neurological repercussions of a FES Cycling session measured by, If sensors present, Intracranial pression.
Cerebral perfusion pressure | During the FES Cycling session (day 1)
  Neurological repercussions of a FES Cycling session measured by, If sensors present, Cerebral perfusion pressure.
Cerebral tissue oxygen pressure | During the FES Cycling session (day 1)
  Neurological repercussions of a FES Cycling session measured by, If sensors present, Cerebral tissue oxygen pressure.
FES cycling installation | After the FES Cycling session (day 1)
  FES Cycling technical feasibility measured by installation and uninstallation times Cycloergometer,
FES Cycling technical feasibility | After the FES Cycling session (day 1)
  FES Cycling technical feasibility measured by number of persons needed.
Duration of FES Cycling session | After the FES Cycling session (day 1)
  FES Cycling technical feasibility measured by total duration of FES Cycling session.
Failure FES Cycling session | After the FES Cycling session (day 1)
  FES Cycling technical feasibility measured by number of procedural failures.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme MOREL, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: Undecided